CLINICAL TRIAL: NCT05786157
Title: Advancing Couple and Family Alcohol Treatment Through Patient-Oriented Research and Mentorship
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Julianne Flanagan, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00127577
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Posttraumatic Stress Disorder; Couples
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will complete an alcohol administration paradigm (peak breath alcohol concentration=.09-.10 g/dL BrAC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- alcohol administration paradigm (Experimental): Participants will complete an alcohol administration paradigm (peak breath alcohol concentration=.09-.10 g/dL BrAC)
  Interventions: Other: Alcohol Administration

INTERVENTIONS:
Other: Alcohol Administration — Participants will complete an alcohol administration paradigm (peak breath alcohol concentration=.09-.10 g/dL BrAC)

SUMMARY:
Intimate partner violence (IPV) is a serious public health problem that results in significant health and economic burdens including mortality, morbidity, and poor treatment outcomes. A well-developed field of research suggests that alcohol misuse and posttraumatic stress disorder (PTSD) can lead to IPV. Individuals with PTSD and/or problematic drinking behaviors are at risk for IPV because of several factors that are common symptoms of PTSD. Because individuals with PTSD often drink alcohol to "self-medicate" or cope with distressing PTSD symptoms, PTSD co-occurs with alcohol misuse and alcohol use disorder at extraordinarily high rates. However, few studies have examined the combined effects of alcohol misuse and PTSD on any form of violence.

This study will examine the effects of alcohol misuse and posttraumatic stress disorder (PTSD) on alcohol-related intimate partner violence (IPV). We will examine these associations among couples (N=70) in a controlled laboratory setting using validated, standardized methods in a 'real-world' settings using 28 days of ecological momentary assessment (EMA).

DETAILED DESCRIPTION:
Alcohol misuse has a salient precipitous effect on intimate partner violence (IPV), which is a persistent public health crisis affecting approximately one-third of the U.S. population. Posttraumatic stress disorder (PTSD) is highly prevalent, has a clear causal effect on alcohol misuse, and it is a robust independent predictor of IPV. However, few studies have examined the combined effects of PTSD and alcohol misuse on IPV. This question is critical to address because effective prevention and treatment approaches for alcohol-related IPV are scant. Integrating these two siloed areas of the literature can help inform the development of novel, trauma-informed modalities for couples to produce stronger and more sustainable outcomes. Dr. Flanagan is the ideal candidate to advance the clinical science in this area. Under the proposed mid-career development award, she will accelerate her thriving patient-oriented alcohol research program by enhancing her skills with 1) oral alcohol administration, 2) intensive ambulatory assessment, and 3) psychophysiology. She will achieve these goals through expert consultation, didactic training, and implementation of the proposed research project. Her team will examine the combined effects of alcohol misuse and PTSD on alcohol-related IPV among couples (N=70) in both a controlled laboratory setting and in naturalistic settings. The study, which was designed to complement mentees' independent research interests, will also compare outcomes across settings and explore heart rate variability as a physiological mechanism underlying the hypothesized relations. The invaluable protected time and resources provided by this K24 will enable Dr. Flanagan to achieve her primary goal of expanding her mentoring availability and skillset at this pivotal mid-career stage. She will engage a program of didactics and expert coaching to amplify her investment in diversity, equity, and inclusion in mentoring, leadership, and science. Achieving these synergistic objectives will accelerate the science of couple and family alcohol research and set the stage for innovative new dyadic treatments. This award will also ensure that Dr. Flanagan is equipped to support the next generation of enthusiastic new investigators and to ensure the longevity of this vital yet underrepresented area of the alcohol field.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender identity; any race or ethnicity; ages 21 years or older.
2. Must report ≥ 2 heavy drinking episodes in the past 30 days (i.e., 4 or more drinks for women, 5 or more for men in ≤ 2 hours) and consumed a quantity of alcohol that is equal to or greater than the standard dose administered for their weight in the laboratory (assessed via the TimeLine Follow Back,TLFB).
3. At least one instance of physical IPV in the current relationship reported by at least one partner within the couple (assessed by the Conflict Tactics Scale, CTS-2).
4. Participants must agree not to drive or operate machinery for the remainder of the experimental visit day. Transportation will be provided if necessary.
5. One or both partners in half the couples will be required to meet diagnostic criteria for PTSD (assessed by the Clinical Administered Posttraumatic Stress Scale, CAPS-5).

Exclusion Criteria:

1. Possible alcohol or drug use disorder (except caffeine or nicotine) as defined by the Alcohol Use Disorders Identification Test, AUDIT scores >8 or Drug Abuse Screening Test DAST scores >3; meeting Diagnostic and Statistical Manual of Mental Disorders, DSM-5 diagnostic criteria; or having ever sought treatment for alcohol or drug use disorder. Recent recreational drug use (e.g., cannabis) is acceptable.
2. Meeting DSM-5 criteria for a history of or current psychotic or bipolar disorders.
3. Current suicidal or homicidal ideation and intent.
4. History of or current psychiatric or medical condition for which alcohol administration is medically contraindicated.
5. Body weight > 250 lbs (in order to rigorously control alcohol dosing).
6. Use of medications such as lithium, methadone, alpha or beta blockers or cholinergic/ anticholinergic drugs likely to confound normative cardiovascular responding for the psychophysiological component of the project.
7. Pregnancy or breastfeeding.
8. Severe or unilateral partner violence in the past 6 months as measured by the CTS-2

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Laboratory intimate partner aggression | 2 hours
  Taylor aggression paradigm
Naturalistic intimate partner aggression | 28 days
  self-report using ecological momentary assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided